CLINICAL TRIAL: NCT06908447
Title: Voluntary Cold-Water Immersion Effects on Value-Based Choice
Brief Title: Cold Water and Decision-Making
Acronym: CoVa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Prof. Dr., German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CoVa; 01GP2210C (Other Grant/Funding Number: German Federal Ministry of Education and Research)
Record Dates: First submitted 2025-03-18; First posted 2025-04-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Behavior; Stress; Quality of Life; Psychological Wellbeing
Keywords: Decision-Making; Psychology; Stress; Cold-Exposure; Cold-Water Immersion
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold-water immersion (Experimental)
  Interventions: Behavioral: Cold-water immersion
- Warm-water immersion (Control) (Experimental)
  Interventions: Behavioral: Warm-water immersion (Control)

INTERVENTIONS:
Behavioral: Cold-water immersion — Single 10-minute acute full-body head-out single arm-out cold-water immersion at 10-16°C on the experimental day
  Arms: Cold-water immersion
Behavioral: Warm-water immersion (Control) — Single 10-minute acute full-body head-out single arm-out cold-water immersion at 30-36°C on the experimental day
  Arms: Warm-water immersion (Control)

SUMMARY:
The behavioral within-subject cross-over design study "CoVa" aims to investigate the effect of a short-term full-body cold-water immersion vs. warm-water immersion control on value-based choice, psychological well-being, and peripheral physiology.

DETAILED DESCRIPTION:
This randomized within-subject cross-over design behavioral study in cognitive neuroscience will employ an acute peripheral physiological intervention, i.e., a 10-minute full-body cold-water (10-16°C) immersion vs. a control condition (10 min @ 30- 36°C water) on two visits separated by approx. 30 days.

Forty eligible female and male participants will be subject to a head-out full-body cold-water immersion or a warm-water condition (control) on two visits. Participants will perform resting-state and task-based non-invasive electrophysiological recordings of the heart, pulse, respiration, skin conductance, and pupil, will undergo thermographic imaging, pre- and post-immersion blood sampling (4 time points), engage in two computer-based decision-making tasks (reinforcement learning task, risk decision-making task), a brief food choice task, and receive a battery of psychometric questionnaires. The visits are separated by approximately 30 days and do not differ in their timeline except for the primary intervention, i.e., cold vs warm-water immersion, and the medical screening on visit 1.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Consent to participate
* Fluency in German
* Physically and mentally healthy
* BMI 18-30 kg/m2
* Normal day-night rhythm

Exclusion Criteria:

* Raynaud syndrome
* Cold urticaria
* High resting heart rate (>160 beats per minute)
* Acute infection
* Diagnosed current or former illnesses of

  * Brain and mind
  * Heart and blood circulation
  * Gastrointestinal system
  * Endocrine system
  * Other serious past or present medical conditions
* Wearing of medical devices (e.g., pacemaker)
* Fear of blood, needles, or phlebotomy
* Allergies to plasters, gels, and other medical equipment
* Allergies to commercially available liquid meals (e.g., shakes, yfood Labs GmbH)
* Recurrent intake of medication which affect metabolism
* Regular nicotine consumption (e.g., vaping, cigarettes)
* Excessive alcohol consumption (>14 servings/week)
* Recent illegal drug consumption (within 2 weeks prior)
* Strong mental or physical stress
* Excessive exercise (>2 h high-intensity exercise/day)
* Pregnancy or breastfeeding
* Inability to wear skin-exposing swimwear, e.g., for religious reasons
* Affinity for winter swimming, cryotherapy, breathwork (>3 times/year)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Risk propensity | On day 1 and after 30 days
  Risk propensity, i.e., the ratio between risky and non-risky choices for each monetary value as measured in the risk decision-making task in the cold-water vs warm-water condition as described in Liu et al. (2021)
Behavioral range adaptation | On day 1 and after 30 days
  Participants will perform a computer-based reinforcement learning task described in Gueguen et al. (2024) to assess reward sensitivity in different monetary contexts. Behavioral range adaptation, which reflects value range-dependent, relative reward valuation, may be altered if reward processing itself is changed through a potent shift in the physiological state. To test whether reward processing is altered after cold vs warm water exposure, the extent to which range adaptation and reference-point centering occurs will be quantified using computational modeling methods.
Food choice | On day 1 and after 30 days
  Participants will be provided an ad libitum restaurant-like breakfast meal during which they can order various food items (e.g., bread, yogurts, cookies) in the desired amount. The ingested food type, nutritional value, and amount will be quantified to assess food preference after cold vs warm water exposure by linking the consumed food with a standardized food database (German Nutrient Database, Bundeslebensmittelschlüssel).
Heart-rate variability | On day 1 and after 30 days
  Task-based and resting-state heart-rate variability, measured with a three-point electrocardiogram (ECG)
Heart rate | On day 1 and after 30 days
  Task-based and resting-state heart rate, measured with ECG
Respiration rate | On day 1 and after 30 days
  Task-based and resting-state respiration rate, measured via a respiration belt
Relative amplitude of the respiratory signal | On day 1 and after 30 days
  Task-based and resting-state relative respiratory amplitude, measured via a respiratory belt
Event-related skin conductance responses | On day 1 and after 30 days
  Phasic electrodermal activity, measured via electrodermal activity (EDA) electrodes
Tonic skin conductance | On day 1 and after 30 days
  Tonic task-based and resting-state electrodermal activity, measured with EDA electrodes
Pupil dilation | On day 1 and after 30 days
  Task-based and resting-state pupil dilation, measured via eye-tracking
Skin temperature | On day 1 and after 30 days
  Thermographic imaging of the face, full-body, supraclavicular, and scapular area using a thermal camera pre-, during, and post-immersion
Plasma concentration of large neutral amino acids | On day 1 and after 30 days
  Large neutral amino acid (LNAA) plasma concentration will be assessed via blood sampling at 4 time points (pre-immersion to 120 min post-immersion)
Plasma concentration of catecholamines | On day 1 and after 30 days
  Catecholamines via blood sampling at 4 time points (pre-immersion to 120 min post-immersion)
Plasma concentration of cortisol | On day 1 and after 30 days
  Cortisol via blood sampling at 4 time points (pre-immersion to 120 min post-immersion)
Identification of epigenetic markers associated with acute cold exposure | On day 1 and after 30 days
  Epigenetic markers (micro-RNA) via blood sampling at 4 time points (pre-immersion to 120 min post-immersion)
Perceived control | On day 1 and after 30 days
  Psychological changes in perceived control, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating high perceived control.
Perceived freedom | On day 1 and after 30 days
  Psychological changes in perceived freedom, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating high perceived freedom.
Perceived stress | On day 1 and after 30 days
  Psychological changes in perceived stress, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating high perceived stress.
State of flow | On day 1 and after 30 days
  Psychological changes in perceived state of flow, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating a high state of flow.
Self-efficacy | On day 1 and after 30 days
  Psychological changes in self-efficacy, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating high self-efficacy.
Perceived pain | On day 1 and after 30 days
  Psychological changes in perceived pain, measured semi-continuously via self-reports throughout the experimental day. Measures range from 0% (not at all) to 100% (very much) with 100% indicating high perceived pain.
Emotions | On day 1 and after 30 days
  Psychological changes in emotions and their bodily origins, measured via self-reports pre- and post-immersion. Measures will be drawn on a virtual body using an adapted version of the Nummenmaa et al. (2014) emBODY tool with red color indicating increased perception and blue indicating decreased perception.
Positive affect and negative affect questionnaire | On day 1 and after 30 days
  Psychological changes in affect, measured semi-continuously via the Positive Affect Negative Affect (PANAS) questionnaire to be filled out pre- and post-immersion. Measures for each item range from 1 (not at all) to 5 (very much) with 5 indicating the highest feeling perceived at the moment.

SECONDARY OUTCOMES:
Trait autonomy questionnaire | On day 1 and after 30 days
  Trait autonomy is assessed via the Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS). Measures range from 1 (not at all true) to 5 (totally true) with 5 indicating the highest score.
Emotion regulation questionnaire | On day 1 and after 30 days
  Emotion regulation, assessed via the Emotion Regulation Questionnaire (ERQ). Measures range from 1 (not at all true) to 7 (totally true) with 7 indicating the highest score.
Causality orientation questionnaire | On day 1 and after 30 days
  Causality orientation, assessed via the General Causality Orientations Scale (GCOS). Measures range from 1 (very unlikely) to 6 (very likely) with 6 indicating the highest probability of responding as the item describes in the vignette scenario.
Delay discounting questionnaire | On day 1 and after 30 days
  Delay discounting is assessed via the Delay Discounting Test by Kirby. Response options to each item are binary with one option corresponding to an immediate reward (e.g., 14 EUR today) and the second option corresponding to a higher but delayed reward (e.g., 19 EUR in 60 days).
Interoceptive awareness questionnaire | On day 1 and after 30 days
  Interoceptive awareness, assessed via the Multidimensional Assessment of Interoceptive Awareness (MAIA) questionnaire. Measures range from 0 (never) to 5 (always) with 5 indicating the highest response.
Generalized self-efficacy questionnaire | On day 1 and after 30 days
  Generalized self-efficacy, assessed via the Self-Efficacy Scale (SWE). Measures range from "not at all true", "hardly true", "moderately true" and "exactly true". A higher score, indicated by a preference for "exactly true", indicated more self-efficacy.
Trait and state anxiety questionnaire | On day 1 and after 30 days
  Trait and state anxiety, assessed via the State-Trait Anxiety Inventory (STAI-S and STAI-T). State anxiety is assessed on a scale from 1 (not at all) to 8 (very much) with a higher score indicating high state anxiety. Trait anxiety is assessed on a scale from 0 (almost never) to 3 (almost always) with a higher score indicating high trait anxiety.
Well-being questionnaire | On day 1 and after 30 days
  Psychological well-being is assessed via the short version of the Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS). Responses range from "never" to "always" on a 5-point scale with a high score indicating higher mental well-being in the past two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Soyoung Q Park, Prof. Dr., Principal Investigator — German Institute of Human Nutrition Potsdam-Rehbruecke
Locations (1):
- German Institute of Human Nutrition Potsdam-Rehbruecke, Nuthetal, Germany

REFERENCES:
- See also: Abler, B. & Kessler, H. (2011). ERQ. Emotion Regulation Questionnaire [Verfahrensdokumentation aus PSYNDEX Tests-Nr. 9006192 und Fragebogen]. In Leibniz-Zentrum für Psychologische Information und Dokumentation (ZPID) (Hrsg.), Elektronisches Testarchi — https://doi.org/10.23668/psycharchives.402
- See also: Scherhorn, G., Haas, H., Hellenthal, F., & Seibold, S. (1999). Kausalitätsorientierungen. Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). — https://doi.org/10.6102/ZIS173
- See also: Forstmeier, S., & Maercker, A. (2011). Selbstkontrolle im höheren Erwachsenenalter: Eine deutsche Version des Delay Discounting Tests von Kirby. PPmP - Psychotherapie · Psychosomatik · Medizinische Psychologie, 61(06), e19-e33. — https://doi.org/10.1055/s-0031-1277169
- See also: Bornemann, B., Herbert, B. M., Mehling, W. E., & Singer, T. (2015). Differential changes in self-reported aspects of interoceptive awareness through 3 months of contempl tive training. Frontiers in Psychology, 5. — https://doi.org/10.3389/fpsyg.2014.01504
- See also: Jerusalem, M., & Schwarzer, R. (2003). SWE - Skala zur Allgemeinen Selbstwirksamkeitserwartung. ZPID (Leibniz Institute for Psychology) - Open Test Archive. — https://doi.org/10.6102/ZIS242
- See also: Grimm, Jürgen (Hg.) (2009): State-Trait-Anxiety Inventory nach Spielberger. Deutsche Lang- und Kurzversion. - Methodenforum der Universität Wien: MF-Working Paper 2009/02 — https://empcom.univie.ac.at/fileadmin/user_upload/p_empcom/pdfs/Grimm2009_StateTraitAngst_MFWorkPaper2009-02.pdf
- See also: Lang, G., & Bachinger, A. (2017). Validation of the German Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) in a community-based sample of adults in Austria: A bi-factor modelling approach. Journal of Public Health, 25(2), 135-146. — https://doi.org/10.1007/s10389-016-0778-8
- See also: Gueguen, M. C. M., Anlló, H., Bonagura, D., Kong, J., Hafezi, S., Palminteri, S., & Konova, A. B. (2024). Recent Opioid Use Impedes Range Adaptation in Reinforcement Learning in Human Addiction. Biological Psychiatry, 95(10), 974-984. — https://doi.org/10.1016/j.biopsych.2023.12.005
- See also: Liu, L., Artigas, S. O., Ulrich, A., Tardu, J., Mohr, P. N. C., Wilms, B., Koletzko, B., Schmid, S. M., & Park, S. Q. (2021). Eating to dare- Nutrition impacts human risky decision and related brain function. NeuroImage, 233, 117951. — https://doi.org/10.1016/j.neuroimage.2021.117951